CLINICAL TRIAL: NCT06823596
Title: Short-term Addition of Efavirenz to Induce CARD8-mediated Reduction of Persistent Nonsuppressible HIV Viremia in People With High Adherence to ART.
Brief Title: The T Cell Activator of Cell Killing ("TACK") IT ON" STUDY
Acronym: "TACKITON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario HIV Treatment Network (Network); Maple Leaf Research (Other); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Mario Ostrowski, Associate Professor, Depts. of Medicine, Immunology. University of Toronto, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46646
Record Dates: First submitted 2024-12-03; First posted 2025-02-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hiv
Keywords: Tack it on
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — efavirenz

STUDY DESIGN:
Intervention Model Description: Pilot study of an already approved HIV drug (Efavirenz), as an addition to current HIV treatment regimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Addition of Efavirenz in people with high adherence to ART. (Other): Single arm - Participants will be prescribed Efavirenz 600 mg q hs x 2 months starting at baseline visit (visit 2)
  Interventions: Drug: Efavirenz 600mg

INTERVENTIONS:
Drug: Efavirenz 600mg — Efavirenz induces pyroptosis of HIV expressing cells via the CARD8 inflammasome. In contrast to most ART drugs, and in addition to its anti-retroviral effect, EFV also induces intracellular Gag-Pol dimerization and premature HIV protease activation, causing cleavage of the inflammasome protein CARD8. CARD8 activation results in the production of effector molecules that rapidly kill virus-infected cells by pyroptosis. This effect of EFV has been called "TACK" or "T cell activator of cell killing". We aim to harness this effect to reduce residual nonsuppresible viremia (NSV) in people on stable antiretroviral therapy (ART). Participants in this study will receive EFV in addition to their stable ART regimen for two months, during and after which we will monitor plasma HIV RNA and markers of viral persistence and immune activation.
  Other Names: Sustiva; Teva-Efavirenz; Mylan-Efavirenz; Jamp-Efavirenz; Auro-Efavirenz

SUMMARY:
Antiretroviral therapy or ART blocks HIV replication reducing plasma viral loads to undetectable levels but has no effect on persistently infected cells in the body, called the virus reservoir. These cells carry infectious HIV capable of restarting HIV replication if therapy is stopped. The reservoir is so stable forcing people to adhere life-long ART. Over 5% of ART adherent individuals continue to have residual non-suppressive viremia (NSV) detected by clinical assays (40-400 copies/ml). Residual viremia reflects a more persistent reservoir and has the potential for increased morbidity. For eg., persistent expression of HIV proteins contributes to inflammation, and can lead to comorbidities. Recently, a novel way to target this reservoir called "TACK" or "Targeted activator of cell killing" is proposed. TACK compounds only target HIV infected cells and directly kill them by inducing a natural killing program (called the inflammasome). Recently the HIV drug, Efavirenz (EFV), which was used to suppress HIV replication for decades, has now been shown to also be a TACK compound. This pilot study will evaluate the impact of Efavirenz (EFV) in reducing HIV persistence by its ability to be a TACK molecule. So in addition to blocking HIV growth, this compound when added to a current ART regimen can kill HIV infected cells in the test tube. We aim to harness this effect to determine whether the addition of EFV to the current ART regimen in people with NSV can suppress the viremia to undetectable levels by killing those cells. NSV represents the "the tip of the iceberg" of those with bigger reservoirs and represents a challenging clinical scenario in dire need of new diagnostic and therapeutic options.

This pilot study will spark larger clinical trials to advance HIV cure strategies, and will provide new tools to improve the clinical management of people living with HIV.

DETAILED DESCRIPTION:
Background:

Combination antiretroviral therapies (cART) have transformed HIV into a chronic manageable health condition for many PLWH.

Despite potent cART, the vast majority of PLWH have residual of viremia that remains below the limit of detection of current clinical assays of 20 copies/ml plasma but can often be detected by highly sensitive assays. A number of studies report that PLWH compliant with cART, without drug resistance mutations, have ongoing detectable low level viremia (also referred to as nonsuppressible viremia, NSV), usually from 20-400 copies/ml, ranging in frequency from 1 in 250 to 9% and 10%. In Ontario, over the past two years, 11.9% of PLWH had two or more consecutive values of low level viremia (LLV) (personal communication Vanessa Tran, Ontario Public Health labs). Although low level viremia on compliant cART is felt not to reflect treatment failure, there is evidence that it may not be clinically insignificant. Recent studies of large cohorts predict a 2-3 fold chance of virologic failure and increased all cause mortality and non-AIDS events with LLV. White et. al. showed that detectable LLV is due to expansion of clones containing both defective and replication competent virus, that are proliferating likely in response to antigens. Thus, individuals with LLV, likely have very large populations of proliferated clones in their reservoirs. Whether this higher level of daily virus production sustains inflammation and immune activation is poorly understood. Moreover, the clinical short-term significance of these findings is unclear, however, these individuals represent a unique group to further study cure strategies that decrease the reservoir size.

Recent observations, suggest that some NNRTIs (especially efavirenz) could be repurposed to kill these virus-producing cells. The HIV protease enzyme is part of a larger gag-pol protein precursor that is produced as an inactive monomer in the cytoplasm of infected cells after HIV transcription. In order for the HIV protease to be active, it must dimerize, and this dimerization only happens within the virus particle that has budded off the cell, which results in mature, infectious viral particles. It has been shown that some NNRTIs such as efavirenz can induce intracellular Gag-Pol dimerization and premature protease activation in the cytosol prior to budding, which can trigger the CARD8 (Caspase recruitment domain protein 8) inflammasome, resulting in death of HIV-1-producing cells via pyroptosis. This process occurs when the compound binds to the RT domain of the Gag-Pol polyprotein, leading to a conformational change that induces its dimerization within the cell cytoplasm rather than in the virus particle, and the consequent autocatalytic activity of the protease enzyme. Thus EFV can induce Gag-pol dimerization in the cytoplasm, which triggers CARD8 sensing and inflammasome activation Intra-cytoplasmic protease-CARD8 activation would be blocked by the presence of protease inhibitors (eg. indinavir). Preliminary data from the Simonetti lab (one of the co-investigators) using CD4+ T cells from people on cART experiencing non-suppressive, but low level viremia, have shown that micromolar concentrations of efavirenz (EFV) can significantly reduce virus production upon strong T cell activation by CD3/CD28 stimulation, due to CARD8 sensing of HIV protease activity . In other words, these virus infected cells were killed in the presence of EFV during immune activation. In control experiments, with the addition of the protease inhibitor lopinavir, the effect of EFV is completely abrogated. Experiments were conducted with EFV at 5uM, which can be reached in plasma in a large fraction of individuals with the recommended full dose (600mg q.d.). Previous pharmacokinetics studies showed that EFV reaching plasma concentration above the EC50 required for its killing effect (1uM) and reaches even higher concentrations in tissues. Recent work reported NNRTI-like molecules with comparable antiviral activity to EFV but significantly higher potency in inducing dimerization and CARD8-mediated killing. However, such compounds are still in the early stages of pre-clinical investigation and their pharmacokinetic profile and activity in vivo has not been explored. This effect, of killing HIV infected cells by pyroptosis after CARD8 sensing has been termed TACK (targeted activator of cell killing). EFV represents the best TACK molecule to test whether the CARD8-inflammasome can be harnessed as a therapeutic option in people living with HIV on ART EFV is recognized as the most promising and potent FDA approved NNRTI compound for this purpose. In the proposed study, cART intensification with EFV is used to induced CARD8 sensing and not to block viral replication.

Hypothesis:

For PLWH, who are adherent to cART, with no documented resistance to their current cART, or EFV, and who have documented persistent nonsuppressible viremia (NSV), the short-term addition of Efavirenz, as a TACK molecule [targeted activator of cell killing], will reduce plasma HIV-1 RNA viral load.

Primary Endpoint Plasma HIV viremia will be compared at baseline (visit 2) after 8 weeks of EFV. (visit 7) Secondary Endpoints

HIV Viral Reservoirs:

QVOA (replication competent virus outgrowth assay) at baseline and at 2 months of EFV Intact proviral DNA assay at baseline, during and after 2 months of EFV Cell-associated HIV RNA at baseline, during and after 2 months of EFV

Immune Activation:

Markers of immune activation and cell death in plasma (baseline and 2 months):

CRP, LDH, IL-1 beta, TNF, IL-6, gasdermin D, Th1 and Th2 cytokines and chemokines Markers of T cell (CD4 and CD8) activation measured at baseline and 2 months via flow cytometry.

T cell resposnes to HIV proteins at baseline and 2 months.

Study Design:

This is a prospective, non-randomized study wherein each enrolled subject will act as their own control before and after the introduction of two months of Efavirenz as a TACK molecule. The study will be at a single site, at Maple Leaf Clinic at Toronto, Unity Health St. Michael's Hospital, and the University of Toronto. After enrollment, the study duration is 20 weeks. All subjects will be recruited to Maple Leaf Clinic, Toronto. Blood draws will occur at Maple Leaf Clinic. Leukapheresis procedures to more intensively study virus reservoirs and immunity will be optional, and will occur at baseline and 8 weeks. Baseline is defined as time to have baseline blood draws, and/or leukapheresis, and individuals will be started on EFV 600 mg PO once daily for 8 weeks, to start the next day. Participants will be identified prior to the baseline visit at about - 4 weeks prior to baseline to ensure eligibility. We intend to enroll 14 participants. At the -4 weeks visit (visit 1), the study pharmacist will review all concomitant medications, compliance, review current ART regimen and the proposed ART regimen with the addition of full dose EFV. Potential side effect/toxicities -espcially EFV's known but reversible neurological effects - and management of them will be discussed. At this time point, a viral load will be obtained to confirm persistent low level viremia. At baseline, (time 0), if prior VL showed LLV, the following assays will be done: HIV viral load, qVOA, IPDA for HIV reservoir measurements, cell-associated HIV RNA, plasma and T cell markers of immune activation, HIV specific T cell immunity. At baseline instead of a 70cc blood draw, subjects will be offered to participate in leukapheresis (optional) which will provide larger cells numbers to better interrogate the HIV reservoir. Subsequent visits at 1 week (V3), 3 weeks (V4), 5 weeks (V5) and 7 weeks (V6) will follow plasma viral load and reservoirs by IPDA. At 8 weeks (V7), participants will discontinue EFV, and viral load, HIV reservoirs, plasma and cell markers of immune activation and T cell immunity will be assayed. Subjects will be offered leukapheresis (optional) to better characterize HIV reservoir and T cell immune studies. Follow up visits will measure plasma viral loads and reservoirs at weeks 9 (V8), 12 (V9) and 16 (V10). At all visits, participants will be reviewed for potential side-effects/toxicities including neuropsychiatric symptoms, and adherence, and CRF reviewed. Potential side effects will be investigated with blood draws and treated accordingly (for e.g., rash, provide antihistamines, HC cream, +/- discontinue EFV if moderate to severe AE by study physician (C. Kovacs). All visits will take place +/- 3 days of the indicated time point.

Sampling. Blood will be collected using SST/EDTA/ACD tubes for the various assays. At baseline and 8 weeks, if subjects undergo leukapheresis, only one 5 ml tube of blood for viral load will be done instead at those time points. Blood volumes are as follows: screening visit (25 ml), 75 ml at all other visits (if leukapheresis not done). At each visit, assessment is made of EFV side effects, new or continuing medications, including cART regimen, and adherence will be assessed. To ensure immune safety, CD4 counts are done at screening, wk 8 and 16.

Statistical Analysis:

Statistical analyses will be conducted with the support of the Johns Hopkins CFAR Biostatistics and Epidemiology core (BEM) and the CTN; differences between time points across the entire cohort will be compared using the Wilcoxon rank-sum or Kruskal-Wallis test. Within-participant (log-transformed) HIV-1 RNA, DNA, changes between time points will be estimated with participant-specific linear regression models and compared against the null hypothesis of no change using the Wilcoxon signed-rank test. The same approach will be applied to soluble markers of immune activation and inflammation.

EXPECTED RESULTS AND IMPLICATIONS The HIV reservoir fails to decay naturally or using cART. The proposed research will address translational aspects of HIV persistence with immediate implications for clinical care. Harnessing CARD8 inflammasome activation with EFV has the potential to eliminate gag/pol transcriptionally active proviruses as a cause of LLV, which at present has limited therapeutic options, given that current antiretroviral agents do not affect virus expression. Reducing LLV could free clinicians and patients from misguided and potentially harmful attempts at unwarranted regimen switching, anxiety of drug failure or personal risks of transmissions to sexual partners. The potential to lower a significant and treatable cause of newly identified adverse inflammation and chronic immune activation has profound implications for improving incidence and outcomes of preventable concomitant diseases. If these efforts advance with discipline, inflammation marker reduction could be used in the HIV treatment clinical care cascade for the first time. Given that much of the reservoir reflects expansion of infected clones, such a strategy may be able to eliminate these. Recently cure studies have experienced participation hesitancy from communities reluctant to agree to cART interruptions in research. This design could provide safety assurance to volunteers while satisfying investigator requirements for reliance on verifiable signals, such as IPDA and vQOA or reduction of LLV. The goal of TACK therapeutics is two fold: 1) to substantially reduce the reservoir of replication competent viruses; and 2) to reduce ongoing antigenic stimulation from clones of latently infected cells containing transcriptionally active but defective viruses interventions that could convert these individuals to undetectable would be beneficial.

RECRUITMENT A total of 26 participants will be recruited for the study.

ELIGIBILITY:
Inclusion criteria for participants are:

* Ability to provide signed written informed consent; age >18 years
* Documented HIV diagnosis
* Continuous antiretroviral therapy for > 4 years with no issues of adherence
* Taking a stable ART regimen, without the inclusion of a protease inhibitor
* At least 4 HIV viral loads >20 and < 400 copies/ml over the past two years
* No documented resistance to EFV in history, no PI including ritonavir in current ART regimen or during study period
* No evidence of EFV resistance by plasma virus sequencing at screening visit
* Non-pregnant throughout the study period, if female sex
* Good general health as shown by medical history and screening laboratory tests at the screening visit:

  * Hemoglobin ≥ 85 g/L, white blood cell count (WBC) > 3,000 cells/mm3
  * Total lymphocyte count .750 X109/L
  * Platelets = 50 to 550 X109/L
  * Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase < 5 times the institutional upper limit of normal (ULN);
* Willing to undergo either leukapheresis or blood draw at visits 2 and 7 (participants will be given the option to undergo blood draws rather than leukapheresis)
* Ability to add efavirenz to their current ART HIV medication re: avoid drug to drug interactions

Exclusion criteria

There will be no exclusion criteria based on gender/gender identity, ethnoracial composition, language, socioeconomic status, mode of HIV acquisition or sexual orientation/identity. Any participant who requires language interpretation can and will be accommodated for by the participation of translators, either at the patient's choice and/or with the assistance of the translator services provided by local ASO organizations. Exclusion criteria for participants include the following:

* Participants who would have difficulty participating in a trial due to non-compliance
* No active medications / illicit drugs that could adversely affect study compliance
* Currently prescribed and using EFV as part of ongoing ART treatment regimen for HIV suppression
* Currently prescribed a protease inhibitor or pharmacologic booster (cobisistat) as part of current ART regimen
* History of major psychiatric condition that would be adversely affected by efavirenz
* Diagnosed severe cognitive impairment or of strong concern in the judgement of investigators that efavirenz would adversely affect participant
* Documented or suspected history of resistance to any NNRTI including efavirenz, nevirapine or rilpivirine
* History of severe intolerance or documented allergy to efavirenz
* Participants with any of the following abnormal laboratory results at the screening visit:

  * Hemoglobin < 85 g/L
  * Lymphocyte count < .750 X109/L
  * Platelet count < 50 X109/L or > 550 X109/L
  * AST or ALT > 5X the upper limit of normal
  * Creatinine > 250 µmol/L
* Participants with a malignancy or undergoing chemotherapy
* Participants with other significant underlying disease (non-HIV-1) that might impinge upon disease progression or death
* Any concurrent condition requiring the continued use of immunoglobulin, antineoplastic agents, glucocorticoids (other than corticosteroid nasal spray for allergic rhinitis; topical or ophthalmic corticosteroids for acute, uncomplicated dermatitis or conjunctivitis; over the counter medications for acute, uncomplicated dermatitis for treatment period not longer than 14 days) or other immunomodulator medications (other than NSAIDS which will be allowed for any length of time)
* Active drug or alcohol use/dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* Any illness or conditions including acute illnesses that, in the opinion of the investigator, may affect the safety of the participant or the evaluation of any study endpoints
* Any other conditions judged by the investigator that would limit the evaluation of a participant
* Any confirmed or suspected immunosuppressive or immunodeficient state (except HIV infection for Group-3), asplenia, recurrent severe infections and chronic use (more than 14 days) immunosuppressant medication within the past six months (topical steroids are allowed)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in plasma viremia (viral copies/ml) | The change in plasma HIV viremia will be compared at baseline (visit 2) versus after 8 weeks of EFV. (visit 7)
  The change in plasma HIV viremia will be compared at baseline (visit 2) versus after 8 weeks of EFV. (visit 7)

SECONDARY OUTCOMES:
The change in plasma HIV viremia will be compared at baseline (visit 2) after 8 weeks of EFV. (visit 7) and after EFV is discontinued (Visits 8 to 10). | compared at baseline and 8 weeks
  1. IPDA - copies/million cells
  2. infectious units per million (quantitative viral outgrowth assay),
  3. cell-associated RNA (unspliced and polyadenylated RNA);

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ostrowski, MD, Principal Investigator — University of Toronto; Colin Kovacs, MD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Unity Health Toronto -St. Michael's Hospital, Toronto, Ontario
  - Maple Leaf Medical Clinic, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
If ever we decide over the coming months to share data with other researcher, an amendment to the protocol and ICF will be submitted for review to research ethics board.